CLINICAL TRIAL: NCT04231110
Title: Combination Therapy With Fecal Microbiota Transplantation and Vedolizumab for Induction of Ulcerative Colitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1001
Record Dates: First submitted 2020-01-02; First posted 2020-01-18 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMT and vedolizumab (Experimental): People who are initiating vedolizumab per standard of care for ulcerative colitis will also be offered FMT weekly for 6 weeks.
  Interventions: Biological: Fecal microbiota transplantation

INTERVENTIONS:
Biological: Fecal microbiota transplantation — Use of fecal microbiota transplantation enemas once weekly in patients who are initiating vedolizumab treatment

SUMMARY:
This is a pilot study of combination therapy using FMT and vedolizumab for induction of UC. The investigators hypothesize that a combination therapy approach which addresses immune trafficking and microbial manipulation simultaneously will lead to superior outcomes than those seen with single agent therapy.

DETAILED DESCRIPTION:
This is a prospective pilot trial involving a single centre (McMaster University Medical Centre) recruiting patients from Hamilton, Ontario Canada and the surrounding regions, to evaluate efficacy and safety outcomes when using fecal microbiota transplantation once weekly for six weeks in UC patients who are initiated on vedolizumab.

A lead in study will be conducted with the first five patients to ensure engraftment of FMT within the colon. Interim analysis will be conducted after these five patients to ensure engraftment within the colon. Data Safety and Monitoring Board will also be informed of the results after the first five patients, including any adverse events. Decision will be made based on these results whether to proceed with the prospective study using FMT weekly for six weeks, or whether to modify the dose/frequency of FMT treatment.

As patients with previous biologic failure tend to have sub-optimal response to vedolizumab monotherapy, this pilot study will focus on recruitment of previous biologic failure patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 or over
2. Active UC defined as total Mayo score of 6 or more points, with endoscopic subscore at > 2
3. Clinician initiating vedolizumab for patients as per standard of care for UC
4. Patient previously has been exposed to one or more biologic or advanced therapies (anti-TNF, JAK inhibitor, anti-interleukin) and never previously exposed to vedolizumab or other anti-integrin therapy.
5. Females of child bearing potential must be willing and able to use acceptable contraception as per Appendix III. II. b. Toxicity section of the Health Canada Guidance

Exclusion Criteria:

1. Participating in another clinical trial
2. Unable to give informed consent
3. Severe comorbid medical illness
4. Concomitant Clostridium difficile infection
5. Increase in medical therapy for UC in the last 4 weeks. Continued treatment with 5-ASA, azathioprine, or 6-mercaptopurine will be permitted if taken at stable dose for ≥4 weeks prior to study entry. Stable dose (same dose for at least 2 weeks) or a tapering dose of steroids will also be permitted provided the dose of steroid is not increased again. Stable intake of probiotic therapy also permitted.
6. New antibiotic therapy in the last 28 days.
7. Dose of infliximab or golimumab in prior four weeks, adalimumab in prior two weeks, or tofacitinib in prior one week.
8. Pregnant women.
9. Clinically significant lactose intolerance
10. Any condition, in the opinion of the investigator, that the treatment may pose a health risk to the subject, based on lab study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Clinical remission | Week 6
  The primary outcome of this pilot trial is rate of remission of UC, defined as a total Mayo score of 2 or less, with no subscore greater than 1, and endoscopic healing with a endoscopic subscore of 0 or 1.

SECONDARY OUTCOMES:
Compliance | Week 6
  Evaluate the number of patients who complete all their FMT and vedolizumab induction visits
Clinical response | Week 6
  Evaluation of fecal microbiota transplant and vedolizumab for rate of clinical response (defined as reduction of Mayo score of 2 or more points) at the end of the trial.
Endoscopic improvement | Week 6
  Evaluation of fecal microbiota transplant and vedolizumab at rate of endoscopic improvement (defined as reduction of endoscopic Mayo score of 1 or more) at the end of the trial.
Fecal microbiome | Week 6
  Compare the fecal microbiome in UC patients in remission versus still active at the end of the trial.
Mucosal microbiome | Week 6
  Compare the mucosal microbiome in UC patients in remission versus still active at the end of the trial.
Adverse events | Week 6
  Qualitative evaluation of adverse events in patients receiving fecal microbiota transplant and vedolizumab

CONTACTS AND LOCATIONS:
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No